CLINICAL TRIAL: NCT04256148
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Study of ALXN1830 in Patients With Warm Autoimmune Hemolytic Anemia
Brief Title: ALXN1830 in Patients With Warm Autoimmune Hemolytic Anemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is withdrawn due to the global impact of the COVID-19 pandemic.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALXN1830-WAI-201
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Warm Autoimmune Hemolytic Anemia
Keywords: Warm autoimmune hemolytic anemia; WAIHA; Immunoglobulin G (IgG)-mediated autoimmune disorder; Pathogenesis
MeSH Terms: interventions — orilanolimab

STUDY DESIGN:
Intervention Model Description: Participants randomized in 1:1:1:1 ratio to 1 of 4 study arms.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ALXN1830 Dosing Regimen 1 (Experimental)
  Interventions: Biological: ALXN1830
- ALXN1830 Dosing Regimen 2 (Experimental)
  Interventions: Biological: ALXN1830
- ALXN1830 Dosing Regimen 3 (Experimental)
  Interventions: Biological: ALXN1830
- Placebo (Active Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ALXN1830 — Administered via intravenous (IV) infusion
  Other Names: SYNT001
  Arms: ALXN1830 Dosing Regimen 1; ALXN1830 Dosing Regimen 2; ALXN1830 Dosing Regimen 3
Other: Placebo — Matching placebo (sterile liquid diluent) administered via IV infusion
  Arms: Placebo

SUMMARY:
The main objective of the study is to evaluate the safety and efficacy of ALXN1830 compared to placebo in adult participants with warm autoimmune hemolytic anemia (WAIHA).

DETAILED DESCRIPTION:
This study will consist of a 4-week Screening period, 13-week Primary Treatment period, and optional Extended Treatment period (up to 2 years).

ELIGIBILITY:
Key Inclusion Criteria:

* Primary or secondary WAIHA, diagnosed at least 6 weeks prior to Screening
* Failed or not tolerated at least 1 prior WAIHA treatment regimen, for example, corticosteroids, rituximab, azathioprine, cyclophosphamide, cyclosporine, mycophenolate mofetil, danazol, or vincristine
* Hemoglobin < 10 g/dL and ≥ 6 g/dL
* Positive direct antiglobulin test (Coombs) (IgG positive, complement C3 [C3] positive or negative)
* Evidence of active hemolysis including any of the following: a) Lactate dehydrogenase (LDH) > upper limit of normal (ULN), b) Haptoglobin < lower limit of normal (LLN), c) Indirect bilirubin > ULN
* Total IgG > 500 mg/dL

Key Exclusion Criteria:

* Human immunodeficiency virus (HIV) infection (positive HIV-1 or HIV-2 antibody test)
* Positive hepatitis B surface antigen (HBsAg) or hepatitis C antibody test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage Of Participants With ≥ 2 Grams (g)/Deciliter (dL) Increase In Hemoglobin (Hgb) From Baseline | Baseline (Day 1) through Day 92

SECONDARY OUTCOMES:
Total Number Of Units Of Packed Red Blood Cells (pRBCs) Transfused | Day 15 through Day 92
Mean Change From Baseline To Day 92 In Quality Of Life, Assessed Via EuroQoL 5 Dimension 5 Level (EQ-5D-5L) Questionnaire | Baseline, Day 92
Mean Change From Baseline To Day 92 In Quality Of Life, Assessed Via Functional Assessment Of Cancer Therapy Anemia (FACT-AN) Questionnaire | Baseline, Day 92
Number Of Weekly Hgb Measurements With Change From Baseline ≥ 2 g/dL | Day 1 through Day 92
Number Of Participants Needing New WAIHA Rescue Medication Or Increase In Dose Of WAIHA Medication | Day 15 through Day 92

CONTACTS AND LOCATIONS:
Locations (1):
- Alexion Study Site, Whittier, California, United States

IPD SHARING:
Plan to Share IPD: No